CLINICAL TRIAL: NCT07176481
Title: Parents Taking Action to Improve Autism Services Access for Navajo Families in Northern Arizona: Intervention Adaptation and Pilot Trial
Brief Title: Diné Parents Taking Action Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: Mercy Care (Unknown)
Responsible Party: Principal Investigator, Olivia Lindly, Associate Professor - Department of Health Sciences, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1620944
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder (ASD); Developmental Disability
Keywords: Autism Spectrum Disorder (ASD); Parent Training Program; Navajo/Diné
MeSH Terms: conditions — Autism Spectrum Disorder; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two groups: immediate intervention or a waitlist control group (intervention later).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Group (Experimental): Participants in this arm will begin the adapted parent training program right away. The program is delivered by trained Navajo Family Advisors who are parents of older children with autism spectrum disorder (ASD). Parents/guardians of children ages 2-12 years with ASD or related developmental concerns will take part in group sessions that focus on learning and practicing evidence-based strategies to support their child's development and family well-being.
  Interventions: Behavioral: Diné Parents Taking Action Program
- Waitlist Control Group (No Intervention): Participants in this arm will be placed on a waitlist and will not begin the program during the initial study period. After the waiting period, they will be offered the adapted parent training program delivered by trained Navajo Family Advisors.

INTERVENTIONS:
Behavioral: Diné Parents Taking Action Program — A culturally adapted parent training program delivered by trained Navajo Family Advisors, focused on teaching parents/guardians evidence-based strategies to support their child's development and family well-being.
  Arms: Immediate Group

SUMMARY:
The goal of this clinical trial is to learn if a family support program helps Navajo parents and guardians of children with autism spectrum disorder (ASD) or other developmental concerns. The main questions it aims to answer are:

* Is the program something families find useful and easy to take part in?
* Does the program raise parents' knowledge and confidence in using strategies that support their child's development?
* Does the program help children improve in areas such as social communication?

Researchers will compare two groups:

* One group of parents will join the program right away.
* The other group will join the program after waiting.

Participants will:

* Be randomly placed into the "immediate" or "waitlist control" group using simple randomization.
* Take part in sessions led by trained Navajo Family Advisors, who are parents of children with ASD.
* Learn and practice strategies they can use at home to support their child
* Answer surveys about their experience, knowledge, and their child's progress

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian of a child between 2 and 12 years of age.
* Child received a diagnosis of autism spectrum disorder (ASD) OR a developmental disability.
* Parent/guardian identifies as Navajo/Diné.

Exclusion Criteria:

* Parent/guardian is 17 years or younger.
* Child is 13 years or older.
* Child did not receive an ASD diagnosis or a developmental disability diagnosis.
* Parent/guardian does not identify as Navajo/Diné.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Parent Knowledge of Evidence-Based Strategies | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on a parent-report survey assessing comprehension and confidence using strategies taught in the program.
Child Social Communication | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on the Social Communication Questionnaire (Rutter, Bailey, & Lord, 2003), a parent-report survey assessing their child's social communication skills.
Frequency Using Intervention Strategies | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on a parent-report survey assessing the frequency of use of the learned intervention strategies.
Family Outcomes | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on the Family Outcomes Survey-Revised, a parent-reported measure of their child's strengths, needs, and abilities (Waschl et al., 2021).

SECONDARY OUTCOMES:
Child problem behavior | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on the Nisonger Child Behavior Rating Form, an assessment of problematic behavior in children (Aman et al., 1996).
Service Use | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Number and type of services the child has received.
Autism Parenting Stress | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on the Autism Parenting Stress Index (Silva & Schalock, 2012).
Parent Health Literacy | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Mean score on the BRIEF Health Literacy Measure (Sand-Jecklin, & Coyle, 2014).
Parent Depression | Immediate intervention group: Baseline, immediate post-intervention, and 2-months post-intervention. Waitlist intervention group: Baseline, 2-months after baseline, and 2-months after second assessment.
  Parent-reported depressive symptoms using the Center for Epidemiological Studies Depression Scale (CES-D).

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Lindly, Ph.D., M.P.H., Principal Investigator — Northern Arizona University
Locations (1):
- Department of Health Sciences - Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Given the policies from the Navajo Nation Human Research Review Board (NNHRRB), all data will go back and belong to the NNHRRB. Individual participant data will not be shared with other researchers for this study.